CLINICAL TRIAL: NCT07005466
Title: Clinical Study of Bronchoalveolar Lavage Combined With High-throughput Sequencing Technology in the Precise Diagnosis of Immunosuppressive Host Pneumonia
Brief Title: Bronchoalveolar Lavage Combined With High-throughput Sequencing Technology
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-019; 2018CR019 (Registry Identifier: Nanfang Hospital, Southern Medical University)
Record Dates: First submitted 2025-05-26; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Pneumonia
Keywords: Immunosuppressive Host control pneumonia; NGS; pneumonia; Checkpoint inhibitor related pneumonia; Pulmonary aspergillosis
MeSH Terms: conditions — Pneumonia; Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Alveolar lavage fluid, venous blood and sputum were collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with lung infections: the positive of CMT or NGS
- Patients without lung infections: the negative of CMT or NGS

SUMMARY:
High-throughput sequencing technology/Metagenomic next generation sequencing (mNGS) has extensive applications in fields such as whole-genome sequencing, transcriptome, gene expression regulation, and epigenetics. Because mNGS has the characteristics of large sequencing throughput, short time and high sensitivity, it can detect thousands of pathogens including bacteria, viruses, true bacteria and parasites, and is widely used in infectious diseases. In 2020, the "Expert Consensus on the Clinical Application of Metagenomic Second-Generation Sequencing Technology in Detecting Infectious Pathogens in China" proposed that for immunodeficient patients, mNGS can significantly increase the detection rate of pathogens and can be used as a first-line detection method. However, at present, there is no unified standard for the interpretation of mNGS results in the environment with bacteria in the respiratory tract, and there are not many studies on the efficacy of mNGS applied in the detection of bacteria and fungi. This study explored the clinical application value of mNGS in the pathogen detection of pneumonia in immunosuppressed hosts.

DETAILED DESCRIPTION:
Infection is the most common complication in immunosuppressed hosts, and lung infection is one of the leading causes of hospitalization and death in immunosuppressed hosts, and accurate pathogenetic diagnosis of pneumonia in immunosuppressed hosts remains challenging at present. Bronchoalveolar lavage is the standard method for sampling microorganisms in the lower respiratory tract, and with the progressive application of high-throughput sequencing (NGS) technology for pathogenetic testing and its success, we have clinically observed that bronchoalveolar lavage combined with NGS improves the rate of pathogenic diagnosis of pneumonia in the immunosuppressed host and benefits the patient. In this project, we plan to prospectively enroll patients with immunosuppressed host pneumonia and perform both bronchoalveolar lavage NGS and clinical conventional sputum culture, blood culture, TB-DNA test, fungal GM test, viral PCR test and other pathogenicity tests, and based on the above results, we will explore whether bronchoalveolar lavage in combination with NGS can increase the rate of pathogenic diagnosis of immunosuppressed host pneumonia and evaluate the effectiveness of the clinical value of NGS in serving as a tool for pneumonia detection and control and in optimizing antibiotic treatment strategies for pneumonia in immunosuppressed hosts.

This study compared the positive rate and accuracy rate of pathogen detection in immunosuppressive host pneumonia by mNGS and CMT, and explored the clinical value of bronchoalveolar lavage combined with high-throughput sequencing technology in the precise diagnosis of immunosuppressive host pneumonia. To increase the etiological diagnosis rate of pneumonia in immunosuppressed hosts, shorten the diagnosis time and improve its prognosis.

ELIGIBILITY:
Inclusion criteria:

1. Voluntary signing of informed consent;
2. Age 14-75 years, No gender limitation；
3. Immunosuppressed host；
4. Symptoms，signs or imaging findings of pneumonia，and ineffective empirical anti-infection treatment；
5. Specimens collected for NGS testing.

Exclusion criteria：

1. No paired conventional microbiological tests (smear，culture，etc.)；
2. Incomplete case records；
3. Inability to complete bronchoalveolar lavage (BAL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet all of the following criteria are eligible to participate in the study:
  Sign the informed consent form voluntarily; Age 18-75 years old, no gender limitation; Immunosuppressive host; Symptoms, signs, or imaging of pneumonia show signs of pneumonia, and empiric anti-infection treatment is ineffective.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity in pneumonia patients | 2021.01-2024.12
  Sensitivity: the ratio of the number of positive cases detected within the experimental group diagnosed with the disease by the gold standard.
  Specificity: the ratio of the number of negative cases detected in the control group diagnosed as disease-free by the gold standard.
Positive predictive value (PPV), negative predictive value (NPV) in pneumonia patients | 2021.01-2024.12
  Positive predictive value: the proportion of positive diagnostic test results to be evaluated that are actually diseased, i.e., the percentage of positive results that are predictive of actual disease.
  Negative predictive value: the proportion of cases that are positive for a given disease among the diagnostic tests to be evaluated, i.e., the percentage of cases that can be predicted to be truly diseased from the positive results.

SECONDARY OUTCOMES:
Therapeutic success rate | 2021.01-2024.12
  Therapeutic success rate: the proportion of cases in which the diagnostic test to be evaluated was positive that were successfully treated.
the proportion of cases in which an adverse event occurs. | 2021.01-2024.12
  Safety: the proportion of cases in which an adverse event occurs.
the average length of stay of patients in the hospital. | 2021.01-2024.12
  Mean length of stay: the average length of stay of patients in the hospital.
Survival rate | 2021.01-2024.12
  Survival rate: the proportion of treated patients who are alive at 30, 60 and 90 days after the onset of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Laiyu, professor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Guangdong Locations, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No